CLINICAL TRIAL: NCT05256602
Title: Prevalence of Knowledge, Attitudes and Perception of Covid Vaccine in Iraq. A Cross Sectional Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: AlFayhaa General Hospital (Other)
Collaborators: University of Basra (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20222
Record Dates: First submitted 2022-02-24; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: COVID-19; Sars-CoV-2 Infection; COVID-19 Pandemic
Keywords: Vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- survey respondant

SUMMARY:
Numerous scientific agencies and iraqi MOH has advised to promote population vaccination as an attempt to reduce the burden of COVID19. The aim of our study is to evaluate knowledge, Attitude, practice and concerns toward different type of covid19 vaccine of Iraqi population. This will help us concentrate our efforts to increase Willingness of vaccination among southren Iraqi people

DETAILED DESCRIPTION:
Detailed Description: New human pandemic disease that have large of world population concern and have many challenges that effect on their life directly or indirectly is coronavirus infection (COVID 19).Numerous scientific agencies and iraqi MOH has advised to promote population vaccination as an attempt to reduce the burden of COVID19 so need to evalute knowledge, Attitude, practice and concerns toward different type of covid19 vaccine of iraqi population to increase willing of vaccination among southren Iraqi population to reduce mortality rate of covid19 and searching for incidence vaccination against it. So to decrease complication of covid19 pandemic, they introduced covid19 vaccine that has essential role to maintain our life. So many companies of manufacturing of covid19 vaccine with different ways by using part of viruses spike of protein or whole virus after attenuated but some Iraqi population hesitancy that delay of acceptance in spite of this vaccination is represent one of method to protect themselves from infected with covid19 in addition attended social event ,shaking hands ,leaving place when talking with other person and still wearing of mask.

Important recognition key for prevention and maintain our life is attitude judgment and how to do this to give positive or negative idea about covid19vaccine according to different source of information that concerning like social media ,experience of previous personal , governmental information and health care professional sources Considering lake of studies and research related to covid19 vaccine in Iraq ,so there is urgent need to know refused or hesitant attitude in southern Iraqi population

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate in the study
* Living in southern Iraq

Exclusion Criteria:

* Less than18 years
* Not willing to complete the questionnaire
* Unable to complete the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults above 18 years old living in southern Iraq.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-03-07 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
KAPC knowledge, Attitude, Practice and Concerns questionnaire | at the time of survey and upto 2 months
  How vaccination and other attitudes are affected by COVID

SECONDARY OUTCOMES:
Factors associated with participants refusing the vaccination | at the time of survey and upto 2 months

IPD SHARING:
Plan to Share IPD: Yes
IPD can be shared with a suitable request from other researchers
Supporting Information: Study Protocol, SAP